CLINICAL TRIAL: NCT03661541
Title: A Phase I Study of the Immune Response to Herpes Simplex Virus Type 1 (HSV-1) and General Immune Health in Subjects Infected With HSV-1
Brief Title: Immune Response and General Immune Health in Subjects Infected With Herpes Simplex Virus Type 1 (HSV-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Squarex, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2017-SQ-Prism
Record Dates: First submitted 2018-05-01; First posted 2018-09-07 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HSV; Herpes Labialis
Keywords: Squaric Acid; Squaric acid dibutyl ester; cold sores
MeSH Terms: conditions — Herpes Labialis | interventions — squaric acid dibutyl ester

STUDY DESIGN:
Intervention Model Description: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  x Group A: 12 subjects with 6 or more herpes labialis outbreaks in the past 12 months x Group B: 12 subjects with 1 to 2 outbreaks in the past 12 months x Group C: 12 subjects with zero outbreaks in the past 12 months Subjects in group A will receive 2% SADBE dose on the arm after their initial blood samples are obtained. Group A subjects will have blood collected and tests repeated 2 and 8 weeks later.
  Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A, 6 or more outbreaks per 12 months (Experimental): Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group A: 12 subjects with 6 or more herpes labialis outbreaks in the past 12 months.
  Subjects in group A will receive 2% Squaric Acid Dibutyl Ester (SADBE) dose on the arm after their initial blood samples are obtained. Group A subjects will have blood collected and tests repeated 2 and 8 weeks later.
  Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
  Interventions: Drug: Squaric Acid Dibutyl Ester
- Group B, 1 or 2 outbreaks per 12 months (No Intervention): Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group B: 12 subjects with 1 to 2 outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Invite these back for a further blood draw on Day 0.
- Group C, zero outbreaks per 12 months (No Intervention): Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group C: 12 subjects with zero outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Invite these back for a further blood draw on Day 0.

INTERVENTIONS:
Drug: Squaric Acid Dibutyl Ester — 2% squaric acid dibutyl ester (SADBE) (Supplied by Squarex) is topically applied to the inner aspect of the upper arm of the subject and covered with Tegaderm. Subject is advised to wash it off after 3 hours.
  Other Names: SADBE
  Arms: Group A, 6 or more outbreaks per 12 months

SUMMARY:
Subjects were recruited who were positive for antibody against herpes simplex virus type 1 (HSV-1) and self-reported having in the previous 12 months

* 6 or more herpes labialis outbreaks (group A),
* 1 or 2 outbreaks (group B), or
* zero outbreaks (group C). Twelve subjects in each group were recruited. Blood was collected from these persons and peripheral blood mononuclear cells (PBMCs) isolated and tested for proliferation in vitro when stimulated with HSV-1-infected cell extracts, free HSV-1 virus, or Candida albicans extract. Candida albicans is a ubiquitous infectious fungus and its extract is used as a test of general immune response. RNA was also isolated from the PBMCs after incubation in the three stimuli and expression of 41 immune-related genes quantified by quantitative real-time PCR. Also serum anti-HSV-1 IgG levels were quantified.

After the blood collection on day 1, the persons in group A (frequent cold sore sufferers) were treated with a single topical application of 2% squaric acid dibutyl ester (SADBE) in DMSO, applied to the inner aspect of the upper arm. These subjects returned on days 15 and 57 for blood collection, and their PBMCs were tested again on those dates for proliferation in vitro against the same stimuli and for gene expression and for serum anti-HSV-1 IgG levels.

DETAILED DESCRIPTION:
Primary oral infection with the herpes simplex virus (HSV) typically occurs at a young age, is asymptomatic, and is not associated with significant morbidity. After primary oral infection, HSV may persist in a latent state in the trigeminal ganglion and later reactivate as the more common herpes labialis, or "cold sores." Common triggers for reactivation are well known and include ultraviolet light, trauma, fatigue, stress, fever, inflammation, and menstruation. These lesions affect up to 45 percent of the U.S. population. They classically manifest as a well-localized cluster of small vesicles along the vermilion border of the lip or adjacent skin. The vesicles subsequently rupture, ulcerate, and crust within 24 to 48 hours. Spontaneous healing occurs over seven to 10 days. In immunocompetent patients, herpes labialis usually is mild and self-limited. However, pain, swelling, and cosmetic concerns may prompt physician consultation. Orally administered antiviral agents, such as acyclovir (Zovirax) or valacyclovir (Valtrex), have a modest clinical benefit if initiated during the prodrome. Topical treatment with 1% penciclovir cream (Denavir) may reduce healing time and pain slightly, even if initiated after the prodrome. However, reduction in healing time with systemic or topical agents is modest. Squaric acid dibutyl ester (SADBE) is a topical immunotherapeutic agent used in the treatment of verruca vulgaris and alopecia areata. During a recent FDA Compounding Advisory Committee Meeting, it was recommended that squaric acid dibutylester be included on the list of bulk drug substances allowed for use in compounding under section 503A of the Federal Food, Drug, and Cosmetic Act. And SADBE has now been so listed under section 503A. A study completed by Lee et al of 29 patients with recalcitrant warts demonstrated complete clearance in 69% of patients with application every 2-4 weeks. Silverberg et al showed a complete clearance in 58% of patients (n=61) when SADBE was applied 3 times weekly. SADBE has also been used with some success in the treatment of alopecia areata. In a review of the literature, Rokhsar et al noted a 50% to 60% success rate of SADBE in use for hair re-growth in this population. SADBE has been reported to cause eczema, lymphadenopathy, blistering, allergic contact dermatitis, skin hypopigmentation, a burning sensation after application, and systemic reactions including fever and arthralgias. A study completed by Oglio et al of eight patients treated with SADBE for warts noted only mild and well tolerated side effects of erythema, desquamation, cutaneous edema, pruritus, burning, and pain. SADBE induces a delayed-type hypersensitivity response which in warts, is believed to induce the killing of virally infected cells by cytotoxic lymphocytes. This influx of lymphocytes into lesional Page 4 of 14 tissue may also enhance the recognition and processing of viral antigens, leading to clonal expansion of effector cells. It is hoped that SADBE will offer subjects a safe and effective therapeutic option to decrease the frequency and severity of future herpes labialis outbreaks through these mechanisms. A placebo-controlled clinical study completed at Massachusetts General Hospital showed that squaric acid prevented recurrence of herpetic lesions. The effect of SADBE of delaying new herpes labialis outbreaks was highly significant (p<0.01) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <65
2. Positive test for IgG against herpes simplex virus type 1 (HSV-1).
3. Groups A and B only: Clinical diagnosis of herpes labialis, which may be made at the screening visit based on the patient's self-reported history of symptoms. An active herpes labialis outbreak at the time of entry into the clinical trial will neither be required nor will be an exclusion criteria.
4. Group A only: Self report having six or more episodes of herpes labialis in the past 12 months. Subjects will NOT be told that six-or-more episodes in the previous 12 months is the entry criterion. Subjects will be asked "How many separate episodes of cold sores have you had in the previous 12 months?" They will be included if they give an answer of six or more and excluded from Group A if they give an answer of five or fewer.
5. Group A only: At least half of the subject's episodes of the previous 12 months should be vesicular in nature and at least half preceded by prodromal symptoms.
6. Group B only: Self report having exactly 1 or 2 episodes of herpes labialis in the past 12 months. Subjects will NOT be told that one or two episodes in the previous 12 months is the entry criterion. Subjects will be asked "How many separate episodes of cold sores have you had in the previous 12 months?" They will be included if they give an answer of one or two and excluded from Group B if they give a different answer.
7. Group C only: Self report having zero episodes of herpes labialis in the past 12 months. Subjects will NOT be told that zero episodes in the previous 12 months is the entry criterion. Subjects will be asked "How many separate episodes of cold sores have you had in the previous 12 months?" They will be included if they give an answer of zero and excluded from Group C if they give an answer of one or more.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Current or recurrent non-herpetic infection or any underlying condition that may predispose to infection or anyone who has been admitted to the hospital due to bacteremia, pneumonia or any other serious infection in the last 12 months.
3. Therapy with glucocorticoid or immunosuppressants at time of recruitment or within past 4 weeks prior to the screening visit (including inhaled corticosteroids for asthma), except for topical steroids in sites other than face.
4. History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers).
5. History of organ transplantation.
6. HIV-positive status determined by history at screening or known history of any other immunosuppressive disease.
7. Severe co-morbidities (diabetes mellitus requiring insulin, CHF (NYHA class II or worse) MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease
8. Known hypersensitivity to Dimethyl sulfoxide (DMSO).
9. Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.
10. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
11. Previous exposure to SADBE (squaric acid or squaric acid dibutyl ester).
12. Subject has an abnormal skin condition (e.g., acne, eczema, rosacea, psoriasis, albinism, or chronic vesiculo-bullous disorder) that occurs in the area ordinarily affected by herpes labialis.
13. Subject has had a vaccine for either HSV-1 or HSV-2.
14. Group A only: People that have had treatment with anti viral therapy within 2 weeks before sensitization dose of SADBE.
15. Groups B and C only: People that have had treatment with anti-viral therapy any time in the past 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Clinical Research
Locations (1):
- Prism Clinical Research, LLC, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McTavish H, Zerebiec KW, Zeller JC, Shekels LL, Matson MA, Kren BT. Immune characteristics correlating with HSV-1 immune control and effect of squaric acid dibutyl ester on immune characteristics of subjects with frequent herpes labialis episodes. Immun Inflamm Dis. 2019 Mar;7(1):22-40. doi: 10.1002/iid3.241. Epub 2019 Feb 12. PMID 30756512

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 or More Herpes Labialis Outbreaks: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group A: 12 subjects with 6 or more herpes labialis outbreaks in the past 12 months.
  Subjects in group A will receive 2% Squaric Acid Dibutyl Ester (SADBE) dose on the arm after their initial blood samples are obtained. Group A subjects will have blood collected and tests repeated 2 and 8 weeks later.
  Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
  Squaric Acid Dibutyl Ester: 2% squaric acid dibutyl ester (SADBE) (Supplied by Squarex) is topically applied to the inner aspect of the upper arm of the subject and covered with Tegaderm. Subject is advised to wash it off after 3 hours.
- 1 to 2 Herpes Labialis Outbreaks: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group B: 12 subjects with 1 to 2 outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Invite these back for a further blood draw on Day 0.
- Zero Herpes Labialis Outbreaks: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group C: 12 subjects with zero outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Invite these back for a further blood draw on Day 0.
Period: Overall Study
Arm/Group | 6 or More Herpes Labialis Outbreaks | 1 to 2 Herpes Labialis Outbreaks | Zero Herpes Labialis Outbreaks
Started | 12 | 12 | 12
Completed | 10 | 10 | 10
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- 1 or 2 Herpes Labialis Outbreaks: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group B: 12 subjects with 1 to 2 outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Invite these back for a further blood draw on Day 0.
- Total: Total of all reporting groups
Arm/Group | 6 or More Herpes Labialis Outbreaks | 1 or 2 Herpes Labialis Outbreaks | Zero Herpes Labialis Outbreaks | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 51.71 [28.3 to 60.4] | 51.71 [28.1 to 61.1] | 54.30 [32.2 to 60.3] | 52.57 [28.1 to 61.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 26
  Male | 3 | 3 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 11 | 9 | 9 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Absolute Gene Expression of IFNG and IL5 in PBMCs Between 8 Weeks and Baseline
Description: RNA gene expression of interleukin-5 (IL5) and interferon gamma (IFNG) genes in PBMCs exposed in vitro to 4 conditions: no stimulus, HSV-1 virus, HSV-1-infected cell extracts, and Candida albicans extract. Measure is qRT-PCR crossing threshold (Ct), where a lower number is higher gene expression. A lower Ct of 1 is approximately a 2-fold higher expression level of the gene.
Time Frame: Baseline and 8 weeks after baseline (Day 1) +/- 7 days for subjects with less than 6 herpres labialis outbreaks in 12 months, relative to baseline for subjects with 6 or greater herpes labialis outbreaks
Population: Absolute gene expression for Group A on Day 57, Group B on day 1 and Group C on day 1 compared to Group A on Day 1.
Measure: Mean (Standard Deviation); unit: q-RT-PCR crossing threshold cycle (Ct)
Groups:
- Group A: 6 or More Herpes Labialis Outbreaks, Day 1: Group A: 12 subjects positive for Ab against HSV-1 and self-reporting 6 or more herpes labialis outbreaks in the past 12 months.
  Subjects in group A will receive 2% Squaric Acid Dibutyl Ester (SADBE) dose on the arm after their initial blood samples on day 1 are obtained. Group A subjects had blood collected and tests repeated 2 and 8 weeks later.
  Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
  Squaric Acid Dibutyl Ester: 2% squaric acid dibutyl ester (SADBE) (Supplied by Squarex) is topically applied to the inner aspect of the upper arm of the subject and covered with Tegaderm. Subject is advised to wash it off after 3 hours.
- Group B: 1 or 2 Herpes Labialis Outbreaks in Prior 12 Months, Day 1: Group B: Subjects positive for Ab against HSV-1 and self-reporting 1 or 2 herpes labialis outbreaks in the prior 12 months.
  Group B: 12 subjects with 1 to 2 outbreaks in the past 12 months. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges. Results from blood draw on day 1.
- Group C: Zero Herpes Labialis Outbreaks in Prior 12 Months, Day 1: Group C: 12 subjects positive for Ab against HSV-1 nad self-reporting zero herpes labialis outbreaks in the past 12 months. Blood draw is on day 1. Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
- Group A, Day 57. Subjects With 6 or More Outbreaks, 8 Weeks After Single Dose of SADBE.: Group A, day 57. Subjects positive for Ab against HSV-1, self-reporting 6 or more herpes labialis outbreaks in the prior 12 months. Blood was collected on day 57 after a single topical dose of SADBE applied to the upper arm on day 1.
Arm/Group | Group A: 6 or More Herpes Labialis Outbreaks, Day 1 | Group B: 1 or 2 Herpes Labialis Outbreaks in Prior 12 Months, Day 1 | Group C: Zero Herpes Labialis Outbreaks in Prior 12 Months, Day 1 | Group A, Day 57. Subjects With 6 or More Outbreaks, 8 Weeks After Single Dose of SADBE.
Number analyzed (Participants) | 12 | 12 | 12 | 12
q-RT-PCR crossing threshold cycle (Ct)
  IL5 in negative control | 10.073 (0.544) | 11.380 (1.233) | 10.711 (1.274) | 11.431 (1.143)
  IL5 with HSV-1-infected cell extract stimulus | 9.624 (0.666) | 10.983 (0.971) | 10.986 (1.268) | 10.627 (0.810)
  IL5 with HSV-1 virus stimulus | 9.747 (0.697) | 10.736 (0.880) | 10.414 (1.217) | 10.595 (0.957)
  IL5 with Candida stimulus | 10.680 (0.941) | 10.806 (1.093) | 11.051 (1.332) | 10.536 (1.215)
  IFNG in negative control | 10.033 (0.820) | 10.210 (1.320) | 9.729 (1.902) | 9.718 (1.164)
  IFNG in HSV-1-infected cell extracts stimulus | 6.040 (1.681) | 3.898 (1.900) | 4.992 (2.418) | 3.522 (1.600)
  IFNG in HSV-1 stimulus | 7.384 (1.670) | 5.554 (2.650) | 5.789 (1.923) | 3.923 (1.548)
  IFNG in Candida stimulus | 8.421 (2.053) | 6.167 (2.980) | 7.336 (1.957) | 5.327 (2.696)

2. Primary Outcome: Immune Monitoring - PBMC Proliferation
Description: PBMC proliferation in response to 3 stimuli: HSV-1 virus, HSV-1-infected cell extracts, and Candida albicans extract.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percent proliferation
Arm/Group | 6 or More Herpes Labialis Outbreaks | 1 to 2 Herpes Labialis Outbreaks | Zero Herpes Labialis Outbreaks
Number analyzed (Participants) | 12 | 12 | 12
percent proliferation
  HSV-1-infected cell extracts | 16.73 (3.94) | 19.26 (5.57) | 20.19 (4.47)
  HSV-1 virus | 8.26 (1.98) | 11.71 (2.98) | 12.70 (3.05)
  Candida extract | 4.47 (1.53) | 4.85 (1.51) | 7.83 (2.19)
  Normalized all three stimuli | 68.33 (10.42) | 83.21 (13.53) | 99.98 (13.92)

3. Primary Outcome: Immune Monitoring - PBMC Proliferation
Description: PBMC proliferation in response to 3 stimuli: HSV-1 virus, HSV-1-infected cell extracts, and Candida albicans extract.
Time Frame: Day 1 and 8 weeks from Day 1 (Initial visit) +/- 7 days for subjects with 6 or more herpes labalis outbreaks
Population: Only subjects with 6 or more herpes labialis outbreaks were treated, therefore only subjects with 6 or more outbreaks are included in this analysis. This set of data compares them at Day 1, before treatment, and analyzed at 8 weeks from Day 1 treatment. Data were not collected at 8 weeks on the subjects with 1 or 2 outbreaks or with zero outbreaks. Data at day 1 on those groups and the subjects with 6 or more outbreaks is reported in Outcome Measure 2.
Measure: Mean (Standard Error); unit: percent proliferation
Groups:
- 6 or More Herpes Labialis Outbreaks at 8 Weeks; 6 or More Herpes Labialis Outbreaks at Day 1: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group A: 12 subjects with 6 or more herpes labialis outbreaks in the past 12 months.
  Subjects in group A will receive 2% Squaric Acid Dibutyl Ester (SADBE) dose on the arm after their initial blood samples are obtained. Group A subjects will have blood collected and tests repeated 2 and 8 weeks later.
  Subjects in Groups B and C will be matched to the subjects in Group A so that demographic characteristics (i.e., gender distribution, age and weight) are within broadly similar ranges.
  Squaric Acid Dibutyl Ester: 2% squaric acid dibutyl ester (SADBE) (Supplied by Squarex) is topically applied to the inner aspect of the upper arm of the subject and covered with Tegaderm. Subject is advised to wash it off after 3 hours.
Arm/Group | 6 or More Herpes Labialis Outbreaks at 8 Weeks | 6 or More Herpes Labialis Outbreaks at Day 1
Number analyzed (Participants) | 12 | 12
percent proliferation
  HSV-1-infected cell extracts | 16.96 (2.62) | 16.73 (3.94)
  HSV-1 virus | 13.37 (2.38) | 8.26 (1.98)
  Candida extract | 7.35 (2.42) | 4.47 (1.53)
  Normalized all three stimuli | 99.97 (13.11) | 73.75 (11.56)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 8 weeks
Description: Only subjects with 6 or more herpes labialis outbreaks (Group A) were treated and therefore, only this group is included in the adverse event reporting. Subjects in the other two groups were not treated with either drug or placebo, and therefore not at risk of adverse events, and they were not followed for adverse events and no adverse event data was collected for those groups.
Groups:
- 6 or More Herpes Labialis Outbreaks: Subjects will be recruited in three groups, all of whom are infected with HSV-1, as shown by having IgG against HSV-1:
  Group A: 12 subjects with 6 or more herpes labialis outbreaks in the past 12 months.
  Subjects in group A will receive 2% Squaric Acid Dibutyl Ester (SADBE) dose on the arm after their initial blood samples are obtained. Group A subjects will have blood collected and tests repeated 2 and 8 weeks later.
  Group B and C subjects (having 0 or 1 to 2 outbreaks in the prior 12 months) were not treated, and therefore not at risk, and adverse event data was not collected on them.
  Squaric Acid Dibutyl Ester: 2% squaric acid dibutyl ester (SADBE) (Supplied by Squarex) is topically applied to the inner aspect of the upper arm of the subject and covered with Tegaderm. Subject is advised to wash it off after 3 hours.
  Only subjects with 6 or more herpes labialis outbreaks (Group A) were treated and therefore, only this group is included in the adverse event reporting. The patients in the zero outbreaks group and 1 to 2 outbreaks group were not treated with either drug or placebo, and therefore not at risk of adverse events, and they were not followed for adverse events and no adverse event data was collected for those groups. So, again, only subjects in Group A (6 or more outbreaks in the prior 12 months) were treated and thus at risk for adverse events, and adverse event data was collected only for that group.
Arm/Group | 6 or More Herpes Labialis Outbreaks
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 or More Herpes Labialis Outbreaks (N=12)
Local reaction (Skin and subcutaneous tissue disorders) | 2 (2) — Stinging at application site
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03661541/Prot_SAP_000.pdf